CLINICAL TRIAL: NCT02700919
Title: A Phase II, Two-Part, Randomised, Multi-Centre, Multinational, Double-Blind, Placebo-Controlled, Parallel Group Study to Compare the Efficacy and Safety of BCT197 When Added on to Standard of Care for the Treatment of Acute Respiratory Exacerbations of Chronic Obstructive Pulmonary Disease Requiring Hospitalisation in Adults
Brief Title: Efficacy and Safety of BCT197 in Subjects With Acute Respiratory Exacerbations of Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MBCT206
Record Dates: First submitted 2016-02-29; First posted 2016-03-07 (Estimated); Results first posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Regimen 1 (Experimental): Drug: BCT197 Dose 1, Day 1 to Day 5
  Interventions: Drug: BCT197
- Regimen 2 (Experimental): Drug: BCT197 Dose 2, Day 1 to Day 5
  Interventions: Drug: BCT197
- Regimen 3 (Placebo Comparator): Placebo Day 1 to Day 5
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCT197 — Capsules will be taken orally with fluids over a 5 day period after randomization
  Arms: Regimen 1; Regimen 2
Drug: Placebo — Capsules will be taken orally with fluids over a 5 day period after randomization
  Arms: Regimen 3

SUMMARY:
The purpose of this study is to compare the efficacy and safety of BCT197 when added on to standard of care in adult subjects with acute respiratory exacerbations of chronic obstructive pulmonary disease requiring hospitalization. Additionally, the study will characterize the pharmacokinetics of BCT197 in adults with COPD. The total duration of the study will be 26 weeks. Subjects will receive study treatment administration over a period of 5 days after randomization. It is expected that approximately 255 subjects will complete the study and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults
* Presence of an active exacerbation of the ongoing COPD requiring hospitalization for treatment
* Subjects with a documented diagnosis of COPD C or D
* Current smokers or ex-smokers
* A documented history of at least one moderate or severe COPD exacerbation in the 12 months preceding the Screening Visit that required antibiotics and/or systemic corticosteroid.
* Current regular treatment for COPD (for at least 2 months prior to the Screening Visit.

Exclusion Criteria:

* Age less than 40 years old
* Current diagnosis of asthma
* Subjects who have already completed treatment for the current exacerbation of COPD
* Subjects currently requiring intensive care unit (ICU) and/or mechanical ventilation
* Received a course of PDE4, p38 or PDE3/4 inhibitors within their respective defined washout periods.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkin, PhD FRCP, Study Director — Mereo BioPharma
Locations (46):
- United States (3):
  - Mereo Research Site, Michigan City, Indiana
  - Mereo Research Site, Baltimore, Maryland
  - Mereo Research Site, Milwaukee, Wisconsin
- Bulgaria (12):
  - Mereo Research Site, Dupnitsa
  - Mereo Research Site, Gabrovo
  - Mereo Research Site, Kardzhali
  - Mereo Research Site, Kozloduy
  - Mereo Research Site, Kyustendil
  - Mereo Research Site, Lovech
  - Mereo Research Site, Montana
  - Mereo Research Site, Razgrad
  - Mereo Research Site, Rousse
  - Mereo Research Site, Shumen
  - Mereo Research Site, Sliven
  - Mereo Research Site, Sofia
- Czechia (3):
  - Mereo Research Site, Kyjov
  - Mereo Research Site, Mělník
  - Mereo Research Site, Slaný
- Mereo Research Site, Dresden, Germany
- Hungary (6):
  - Mereo Research Site, Balassagyarmat
  - Mereo Research Site, Budapest
  - Mereo Research Site, Debrecen
  - Mereo Research Site, Farkasgyepű
  - Mereo Research Site, Miskolc
  - Mereo Research Site, Mohács
- Mereo Research Site, Naples, Italy
- Latvia (3):
  - Mereo Research Site, Daugavpils
  - Mereo Research Site, Riga
  - Mereo Research Site, Valmiera
- Poland (5):
  - Mereo Research Site, Chrzanów
  - Mereo Research Site, Krakow
  - Mereo Research Site, Proszowice
  - Mereo Research Site, Wroclaw
  - Mereo Research Site, Zgierz
- Romania (7):
  - Mereo Research Site, Bucharest
  - Mereo Research Site, Cluj-Napoca
  - Mereo Research Site, Constanța
  - Mereo Research Site, Craiova
  - Mereo Research Site, Marghita
  - Mereo Research Site, Suceava
  - Mereo Research Site, Timișoara
- Russia (5):
  - Mereo Research Site, Izhevsk
  - Mereo Research Site, Kemerovo
  - Mereo Research Site, Saint Petersburg
  - Mereo Research Site, Saratov
  - Mereo Research Site, Tomsk

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BCT197 High Dose Regimen: Participants received 75 mg BCT197 orally on Day 1. Subsequent doses with 40 mg BCT197 were administered orally on Day 3 and Day 5, respectively. All participants also received standard of care treatment for the acute exacerbation.
- BCT197 Low Dose Regimen: Participants received 40 mg BCT197 orally on Day 1. Subsequent doses with 20 mg BCT197 were administered orally on Day 3 and Day 5, respectively. All participants also received standard of care treatment for the acute exacerbation.
- Placebo: Participants received placebo orally on Day 1. Subsequent doses with placebo were administered orally on Day 3 and Day 5, respectively. All participants also received standard of care treatment for the acute exacerbation.
Period: Overall Study
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Started | 94 | 97 | 91
Completed | 82 | 85 | 87
Not Completed | 12 | 12 | 4
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 1
Not completed — Withdrawal by Subject | 5 | 8 | 2
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Other | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) Population: all randomized patients who received at least one dose of the study medication and who provided a Baseline and at least one post-Baseline forced expiratory volume in one second (FEV1) value.
Groups:
- Total: Total of all reporting groups
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo | Total
Number analyzed (Participants) | 87 | 93 | 86 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.34) | 63.1 (8.68) | 64.7 (7.06) | 63.8 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 26 | 27 | 74
  Male | 66 | 67 | 59 | 192
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 1
  White | 87 | 92 | 85 | 264
  Other | 0 | 0 | 1 | 1
FEV1 at Screening [Mean (Standard Deviation); unit: litre] — Population: Only part of the participants had pre-bronchodilator spirometry results at Screening.
  litre
    Pre-bronchodilator: number analyzed (Participants) | 23 | 25 | 20 | 68
    Pre-bronchodilator | 0.875 (0.3649) | 0.871 (0.3091) | 0.921 (0.2775) | 0.887 (0.3166)
    Post-bronchodilator | 1.135 (0.3875) | 1.046 (0.4009) | 1.033 (0.3558) | 1.071 (0.3836)
Forced Vital Capacity (FVC) at Screening [Mean (Standard Deviation); unit: litre] — Population: Only part of the participants had pre-bronchodilator spirometry results at Screening.
  litre
    Pre-bronchodilator: number analyzed (Participants) | 23 | 25 | 20 | 68
    Pre-bronchodilator | 2.410 (0.8883) | 2.137 (0.8675) | 2.352 (0.7623) | 2.293 (0.8416)
    Post-bronchodilator | 2.619 (0.8167) | 2.514 (0.8488) | 2.427 (0.7298) | 2.521 (0.8022)
FEV1/FVC at Screening [Mean (Standard Deviation); unit: Ratio] — Population: Only part of the participants had pre-bronchodilator spirometry results at Screening.
  Ratio
    Pre-bronchodilator: number analyzed (Participants) | 23 | 25 | 20 | 68
    Pre-bronchodilator | 0.381 (0.1109) | 0.424 (0.0982) | 0.404 (0.0972) | 0.403 (0.1025)
    Post-bronchodilator | 0.447 (0.1245) | 0.427 (0.1107) | 0.436 (0.1184) | 0.436 (0.1177)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in FEV1 to Day 7 - ITT Population
Description: FEV1 data were recorded daily from Days 1 to 7 of the study using a computer-operated spirometer. Analysis was based on a linear Mixed Model for Repeated Measures (MMRM) with Change from Baseline in parameter as outcome; including treatment, visit, treatment by visit interaction, severity of airflow limitation at Baseline, blood eosinophils (%) at Baseline, time from start of current chronic obstructive pulmonary disease (COPD) exacerbation to first study treatment dosing, presence of cardiovascular comorbidities at Screening and COPD exacerbation treatment at Screening as fixed effects, and Baseline value and Baseline by visit interaction as covariates. Baseline was defined as the last non-missing value collected before the first study treatment administration, including unscheduled assessments. Results were presented with adjusted mean (95% confidence interval).
Time Frame: Days 1 to 7
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: litre
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
litre | 0.084 [0.019 to 0.149] | 0.115 [0.049 to 0.180] | 0.057 [-0.011 to 0.125]
Statistical Analysis 1: Comparison: BCT197 High Dose Regimen; Change from Baseline on Day 7; Test type: Superiority; p = 0.012, Log Rank
Statistical Analysis 2: Comparison: BCT197 Low Dose Regimen; Change from Baseline on Day 7; Test type: Superiority; p < 0.001, Log Rank
Statistical Analysis 3: Comparison: Placebo; Change from Baseline on Day 7; Test type: Superiority; p = 0.102, Log Rank
Statistical Analysis 4: Comparison: BCT197 High Dose Regimen vs Placebo; Day 7; Test type: Superiority; p = 0.507, Mixed Models Analysis; Mean Difference (Final Values) = 0.027, 95% CI 2-sided [-0.053 to 0.107]
Statistical Analysis 5: Comparison: BCT197 Low Dose Regimen vs Placebo; Day 7; Test type: Superiority; p = 0.148, Mixed Models Analysis; Mean Difference (Final Values) = 0.058, 95% CI 2-sided [-0.021 to 0.136]
Statistical Analysis 6: Comparison: BCT197 High Dose Regimen vs BCT197 Low Dose Regimen; Day 7; Test type: Superiority; p = 0.443, Mixed Models Analysis; Mean Difference (Final Values) = -0.031, 95% CI 2-sided [-0.109 to 0.048]

2. Secondary Outcome: Change From Baseline in FEV1 on Days 3, 10, and 14 - ITT Population
Description: FEV1 data were recorded daily from Days 1 to 7, and Days 10 and 14 of the study using a computer-operated spirometer. Analysis was based on a linear MMRM with Change from Baseline in parameter as outcome; including treatment, visit, treatment by visit interaction, severity of airflow limitation at Baseline, blood eosinophils (%) at Baseline, time from start of current COPD exacerbation to first study treatment dosing, presence of cardiovascular comorbidities at Screening and COPD exacerbation treatment at Screening as fixed effects, and Baseline value and Baseline by visit interaction as covariates. Baseline was defined as the last non-missing value collected before the first study treatment administration, including unscheduled assessments.
Time Frame: Days 3, 10, and 14
Population: ITT Population
Measure: Mean (Standard Deviation); unit: litre
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
litre
  Day 3: number analyzed (Participants) | 86 | 93 | 84
  Day 3 | 0.026 (0.2118) | 0.059 (0.2101) | 0.063 (0.2392)
  Day 10: number analyzed (Participants) | 82 | 90 | 85
  Day 10 | 0.095 (0.2900) | 0.071 (0.1995) | 0.063 (0.2879)
  Day 14: number analyzed (Participants) | 83 | 88 | 85
  Day 14 | 0.047 (0.2627) | 0.056 (0.2782) | 0.056 (0.2670)

3. Secondary Outcome: Normalization Evaluation of FEV1 Over Time (Days 1 to 7, Days 10 and 14, and Weeks 8, 12 and 26) Compared With the Most Recent Test Performed Within the Last 12 Months Outside an Exacerbation - ITT Population
Description: FEV1 data were recorded daily from Days 1 to 7 and on Days 10 and 14 and Weeks 8, 12, and 26 of the study using a computer-operated spirometer. FEV1 normalization was achieved if FEV1 returned to a value ≥ 89% of the most recent FEV1 value measured within the last 12 months outside an exacerbation (pre-study FEV1 value). Baseline was defined as the last non-missing value collected before the first study treatment administration, including unscheduled assessments. Percentages (%) were based on number of non-missing values as denominator.
Time Frame: Baseline, Days 1 to 7, Days 10 and 14, Week 8, Week 12 and Week 26
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
percentage of participants
  Baseline | 67.9 | 59.3 | 64.6
  Day 2 | 61.9 | 65.2 | 73.2
  Day 3 | 67.5 | 62.6 | 75.0
  Day 4 | 62.7 | 65.9 | 75.0
  Day 5 | 71.1 | 70.2 | 74.7
  Day 6 | 76.8 | 70.5 | 75.0
  Day 7 | 71.6 | 71.6 | 70.4
  Day 10 | 77.2 | 65.9 | 66.7
  Day 14 | 69.1 | 61.6 | 75.3
  Week 8 | 74.0 | 65.4 | 71.4
  Week 12 | 70.5 | 63.0 | 68.8
  Week 26 | 75.7 | 67.1 | 69.3

4. Secondary Outcome: Normalization Evaluation of FEV1/FVC Over Time (Days 1 to 7, Days 10 and 14, and Weeks 8, 12 and 26) Compared With the Most Recent Test Performed Within the Last 12 Months Outside an Exacerbation - ITT Population
Description: FEV1 and FVC were recorded daily from Days 1 to 7 and on Days 10 and 14 and Weeks 8, 12, and 26 of the study using a computer-operated spirometer. FEV1/FVC normalization was achieved if FEV1/FVC returned to a value ≥ 89% of the most recent FEV1/FVC value measured within the last 12 months outside an exacerbation (pre-study FEV1/FVC value). Baseline was defined as the last non-missing value collected before the first study treatment administration, including unscheduled assessments.
Time Frame: Baseline to Week 26
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
percentage of participants
  Baseline | 49.4 | 47.8 | 45.8
  Day 2 | 51.8 | 50.0 | 55.4
  Day 3 | 54.9 | 53.3 | 50.6
  Day 4 | 53.7 | 48.8 | 51.9
  Day 5 | 57.3 | 47.0 | 48.8
  Day 6 | 51.9 | 50.6 | 51.9
  Day 7 | 53.8 | 51.7 | 51.2
  Day 10 | 52.6 | 47.1 | 46.3
  Day 14 | 50.0 | 48.2 | 47.6
  Week 8 | 53.9 | 46.3 | 51.3
  Week 12 | 51.9 | 43.8 | 51.3
  Week 26 | 54.8 | 47.4 | 51.3

5. Secondary Outcome: Time to Improvement of 100 mL in FEV1 Over Time - ITT Population
Description: Time to improvement of 100 mL in FEV1 was defined as time (in days) from initiation of study treatment until the change in FEV1 was ≥ +100 mL.
Time Frame: Baseline to Week 26
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
days | 3.0 [2.0 to 5.0] | 2.0 [2.0 to 4.0] | 4.0 [2.0 to 9.0]
Statistical Analysis 1: Comparison: BCT197 High Dose Regimen vs Placebo; Test type: Superiority; p = 0.399, Log Rank
Statistical Analysis 2: Comparison: BCT197 Low Dose Regimen vs Placebo; Test type: Superiority; p = 0.091, Log Rank
Statistical Analysis 3: Comparison: BCT197 High Dose Regimen vs BCT197 Low Dose Regimen; Test type: Superiority; p = 0.437, Log Rank

6. Secondary Outcome: Area Under the Curve (AUC) of FEV1 Over Time - ITT Population
Description: AUC was calculated according to the trapezoidal rule. The trapezoidal rule is a numerical method to be used to approximate the integral or the area under a curve. Using trapezoidal rule to approximate the area under a curve first involves dividing the area into a number of strips of equal width. Then, approximating the area of each strip by the area of the trapezium formed when the upper end is replaced by a chord. The sum of these approximations gives the final numerical result of the AUC.
Time Frame: Day 1 to Day 14
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mg/(mL*min)
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
mg/(mL*min)
  Day 1-3 | 1.207 (0.4090) | 1.111 (0.4245) | 1.097 (0.3876)
  Day 1-7 | 1.232 (0.4296) | 1.143 (0.4433) | 1.108 (0.3980)
  Day 1-10 | 1.263 (0.4934) | 1.174 (0.4380) | 1.155 (0.4061)
  Day 1-14 | 1.293 (0.4743) | 1.192 (0.4007) | 1.125 (0.4293)

7. Secondary Outcome: Normalization of Respiratory Rate (RR) Over Time During Acute Exacerbation Phase - ITT Population
Description: RR was normalized when it returned to a baseline plateau level achieved after the acute COPD exacerbation during the Stabilization Phase. Baseline was defined as the last non-missing value collected before the first study treatment administration, including unscheduled assessments.
Time Frame: Day 1 to Day 14
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
percentage of participants
  Baseline | 14.9 | 20.4 | 17.4
  Day 2 | 28.7 | 26.9 | 26.7
  Day 3 | 28.7 | 39.8 | 29.4
  Day 4 | 37.9 | 45.1 | 37.6
  Day 5 | 41.4 | 52.7 | 39.3
  Day 6 | 44.8 | 48.4 | 48.2
  Day 7 | 51.2 | 51.6 | 47.1
  Day 10 | 47.6 | 60.4 | 48.2
  Day 14 | 57.8 | 52.3 | 56.5

8. Secondary Outcome: Change From Baseline in RR on Days 3, 7, 10 and 14 - ITT Population
Description: RR (breaths/min) was recorded over time during the acute exacerbation phase.
Time Frame: Days 1 to 14
Population: ITT Population
Measure: Median (Full Range); unit: breaths/min
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
breaths/min
  Day 3: number analyzed (Participants) | 87 | 93 | 85
  Day 3 | -2.0 [-8.0 to 3] | -1.0 [-8.0 to 5.0] | -2.0 [-8.0 to 2.0]
  Day 7: number analyzed (Participants) | 86 | 91 | 85
  Day 7 | -3.0 [-13.0 to 8.0] | -2.0 [-13.0 to 4.0] | -2.0 [-12.0 to 1.0]
  Day 10: number analyzed (Participants) | 84 | 91 | 85
  Day 10 | -3.0 [-13.0 to 4.0] | -2.0 [-14.0 to 4.0] | -2.0 [-12.0 to 2.0]
  Day 14: number analyzed (Participants) | 83 | 88 | 85
  Day 14 | -3.0 [-13.0 to 4.0] | -2.0 [-16.0 to 6.0] | -3.0 [-12.0 to 1.0]

9. Secondary Outcome: Time to Improvement Based on the EXAcerbations of Chronic Pulmonary Disease Tool-Patient Reported Outcome (EXACT-PRO) Total Score During the Acute Exacerbation Phase - ITT Population
Description: Improvement based on EXACT-PRO total score is defined as a decrease in the Rolling Average EXACT score ≥ 9 points from the previous day's maximum observed value during an event. The EXACT is a 14-item patient reported outcome (PRO) daily diary used to quantify and measure exacerbations of COPD. The health status of the participant is correlated to the global score, meaning a higher score corresponds to a more severe health status of the participant. An EXACT Total score is computed for each day of diary collection. The EXACT Total score is based on a logit scoring system with conversion to a 0 to 100 scale for ease of interpretation and use. The total score was used in the determination of exacerbation frequency, severity and duration of exacerbation. Specifically, changes in the total score were used to define onset and recovery from an exacerbation event and the magnitude of that event.
Time Frame: Days 1 to 29
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
days | 5.0 [3.0 to 16.0] | 6.0 [3.0 to NA] — Insufficient data to evaluate the upper limit | 5.0 [3.0 to 7.0]
Statistical Analysis 1: Comparison: BCT197 High Dose Regimen vs Placebo; Test type: Superiority; p = 0.720, Log Rank
Statistical Analysis 2: Comparison: BCT197 Low Dose Regimen vs Placebo; Test type: Superiority; p = 0.298, Log Rank
Statistical Analysis 3: Comparison: BCT197 High Dose Regimen vs BCT197 Low Dose Regimen; Test type: Superiority; p = 0.470, Log Rank

10. Secondary Outcome: Time to Recovery Based on EXACT-PRO Total Score During the Acute Exacerbation Phase - ITT Population
Description: Recovery based on EXACT-PRO total score was defined as the first day in which a participant experiences a persistent, sustained improvement in their condition over the observed period (Day 1 to Day 29). Improvement had to be present for 7 consecutive days. The first day of the 7-day period was designated as the first day of Recovery. An EXACT total score was computed for each day of diary collection.
Time Frame: Days 1 to 29
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
days | 6.0 [NA to NA] — Insufficient data to evaluate the upper and lower limit | 6.0 [NA to NA] — Insufficient data to evaluate upper and lower limit | 6.0 [6.0 to 7.0]

11. Secondary Outcome: Standardized AUC of EXACT-PRO Rolling Average Over Time During Acute Exacerbation Phase - ITT Population
Description: The standardized AUC of the EXACT-PRO were calculated from Day (a) to Day (b) using the trapezoidal rule.
Time Frame: Days 1 to 29
Population: ITT Population
Measure: Median (Full Range); unit: mg/(mL*min)
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
mg/(mL*min)
  Day 1-7: number analyzed (Participants) | 80 | 84 | 82
  Day 1-7 | 45.389 [20.58 to 64.94] | 44.736 [19.61 to 63.19] | 43.938 [19.00 to 67.75]
  Day 1-14: number analyzed (Participants) | 75 | 82 | 81
  Day 1-14 | 42.641 [21.81 to 63.38] | 42.250 [22.80 to 64.87] | 42.590 [17.74 to 65.42]
  Day 1-29: number analyzed (Participants) | 73 | 80 | 80
  Day 1-29 | 41.470 [19.43 to 62.92] | 40.932 [19.81 to 65.25] | 41.652 [20.35 to 61.27]

12. Secondary Outcome: Standardized AUC of EXACT-PRO (Breathlessness) Rolling Average Over Time During Acute Exacerbation Phase - ITT Population
Description: Information regarding the participant's condition can be obtained through 3 domain scores embedded within the EXACT measure: Breathlessness, Cough & Sputum, and Chest Symptoms. These scores also range from 0 to 100 with higher scores indicating more severe symptoms.The standardized AUC of the EXACT-PRO were calculated from Day (a) to Day (b) using the trapezoidal rule.
Time Frame: Days 1 to 29
Population: ITT Population
Measure: Median (Full Range); unit: mg/(mL*min)
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
mg/(mL*min)
  Day 1-7: number analyzed (Participants) | 79 | 83 | 81
  Day 1-7 | 50.083 [21.58 to 80.00] | 47.861 [15.58 to 78.00] | 47.556 [13.13 to 85.50]
  Day 1-14: number analyzed (Participants) | 74 | 81 | 80
  Day 1-14 | 45.417 [21.27 to 79.65] | 45.577 [20.60 to 77.73] | 44.436 [17.41 to 80.69]
  Day 1-29: number analyzed (Participants) | 72 | 78 | 79
  Day 1-29 | 44.911 [23.27 to 79.41] | 45.315 [17.84 to 77.63] | 43.387 [18.65 to 74.91]

13. Secondary Outcome: Rate of Positively Adjudicated Moderate/Severe COPD Exacerbations - ITT Population
Description: Follow-up time per participant (years) was defined as (date of last contact - date of first study drug administration + 1)/ 365.25. Total follow-up time (years) = sum of individual participant follow-up times. Rate was calculated as total number of positively adjudicated exacerbations divided by the total follow-up time in years of the treatment group.
Time Frame: Day 1 to End of Study (Day 180)
Population: ITT Population
Measure: Number; unit: proportion of participants
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
proportion of participants | 0.744 | 0.921 | 0.904

14. Secondary Outcome: Number of COPD-Related Deaths During the Study - ITT Population
Description: Cumulative incidences of COPD-related deaths until Day 30/60/90/120/150/180 were obtained.
Time Frame: Days 1 to 180
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
Participants
  Until Day 30 | 0 | 0 | 1
  Until Day 60 | 0 | 0 | 1
  Until Day 90 | 0 | 0 | 1
  Until Day 120 | 0 | 0 | 1
  Until Day 150 | 1 | 0 | 1
  Until Day 180 | 1 | 0 | 1

15. Secondary Outcome: Time to Next Positively Adjudicated Moderate/Severe COPD Exacerbation- ITT Population
Description: Time to next positively adjudicated moderate/severe COPD exacerbation (in days) was defined as date when first moderate/severe COPD exacerbation symptoms started - date when current COPD exacerbation symptoms stopped, where COPD exacerbations experienced during the study were positively adjudicated by the Independent Adjudication Committee. Time to next positively adjudicated COPD exacerbation was presented in 25th percentile (95% confidence interval) as medians were not evaluable.
Time Frame: Day 1 to Day 180
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
days | 168.0 [70.0 to NA] — Insufficient data to evaluate the upper limit | 75.0 [45.0 to 136.0] | 143.0 [48.0 to NA] — Insufficient data to evaluate the upper limit

16. Secondary Outcome: Time From Hospitalization Admission Until the Participant Is Medically Ready for Discharge (Current COPD) - ITT Population
Description: Time from hospitalization admission until the participant is medically ready for discharge (in days) = Date participant was medically ready for discharge from hospital - Date of hospitalization admission. Date of hospitalization admission' and 'Date participant was medically ready for discharge from hospital' were recorded on the 'Current COPD Exacerbation' form of the eCRF. Results were presented with 75th percentile (95% CI) due to the fact that 95% CI for the median was not evaluable.
Time Frame: Day 1 to Day 30
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
days | 9.0 [8.0 to 12.0] | 9.0 [8.0 to 13.0] | 9.0 [8.0 to 10.0]

17. Secondary Outcome: Percentage of Days With Intake of COPD Rescue Therapy - ITT Population
Description: Participants completed the EXACT-PRO starting from Day 1 and recorded rescue medication use and any occurrences of COPD once a day (evening) in the diary. The percentage of days with intake of rescue medications was evaluated on the basis of the information recorded daily by the participant on the diaries. A day was considered with intake of rescue medications if the answer to the question "How many puffs of rescue medication did you take since last evening?" was> 0.
Time Frame: Baseline to Week 26
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
Number analyzed (Participants) | 87 | 93 | 86
percentage of days
  Acute Exacerbation Phase (Overall) | 73.28 (32.721) | 71.90 (33.565) | 69.65 (35.674)
  Stabilization Phase (Overall): number analyzed (Participants) | 80 | 84 | 83
  Stabilization Phase (Overall) | 70.78 (37.122) | 71.08 (40.299) | 67.35 (38.953)

18. Other Pre Specified Outcome: Pharmacokinetic (PK) of BCT197 in Adults With COPD - PK Population
Description: Descriptive summary of PK plasma concentration is presented as no-specific PK report is available.
Time Frame: Days 1 to 5
Population: PK Population: all participants who received at least one dose administration and had at least one quantifiable plasma concentration.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen
Number analyzed (Participants) | 92 | 92
ng/mL
  Day 1 (0-2 h post-dose): number analyzed (Participants) | 69 | 68
  Day 1 (0-2 h post-dose) | 97.40 [65.13 to 145.66] | 75.98 [47.81 to 120.73]
  Day 1 (4-8h post dose): number analyzed (Participants) | 69 | 68
  Day 1 (4-8h post dose) | 387.65 [343.22 to 437.83] | 283.79 [261.28 to 308.25]
  Day 1 (>12h post-dose): number analyzed (Participants) | 69 | 68
  Day 1 (>12h post-dose) | 413.85 [376.28 to 455.17] | 286.40 [267.20 to 306.97]
  Day 3 (pre-dose): number analyzed (Participants) | 67 | 70
  Day 3 (pre-dose) | 271.10 [251.34 to 292.41] | 161.13 [147.69 to 175.80]
  Day 3 (0-2h post-dose): number analyzed (Participants) | 68 | 70
  Day 3 (0-2h post-dose) | 318.88 [290.57 to 349.95] | 184.46 [165.72 to 205.31]
  Day 3 (4-8h post-dose): number analyzed (Participants) | 68 | 70
  Day 3 (4-8h post-dose) | 496.31 [457.30 to 538.64] | 299.79 [281.99 to 318.71]
  Day 3 (>12h post-dose): number analyzed (Participants) | 68 | 71
  Day 3 (>12h post-dose) | 466.86 [434.70 to 501.40] | 249.60 [231.21 to 269.46]
  Day 5 (pre-dose): number analyzed (Participants) | 39 | 38
  Day 5 (pre-dose) | 272.43 [246.62 to 300.95] | 128.38 [111.99 to 147.17]
  Day 5 (0-2h post-dose): number analyzed (Participants) | 39 | 36
  Day 5 (0-2h post-dose) | 310.20 [277.37 to 346.91] | 155.10 [130.77 to 183.94]
  Day 5 (4-8h post-dose): number analyzed (Participants) | 39 | 36
  Day 5 (4-8h post-dose) | 504.53 [453.33 to 561.52] | 278.73 [246.56 to 315.10]
  Day 5 (>12h post-dose): number analyzed (Participants) | 39 | 36
  Day 5 (>12h post-dose) | 465.28 [423.05 to 511.72] | 240.31 [215.77 to 267.63]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from signing the informed consent form to completion of the 26 week follow-up period after the last administration of study drug.
Description: Serious AEs are also included in the non-serious AE section as a non-serious AE table was not available. The difference in numbers between the participant flow module and safety population is because some participants were randomized but did not go on to receive at least one dose of study medication.
Arm/Group | BCT197 High Dose Regimen | BCT197 Low Dose Regimen | Placebo
All-Cause Mortality (participants affected / at risk) | 2/92 | 3/96 | 2/91
Serious Adverse Events (participants affected / at risk) | 17/92 | 27/96 | 29/91
Other Adverse Events (participants affected / at risk) | 56/92 | 63/96 | 62/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCT197 High Dose Regimen (N=92) | BCT197 Low Dose Regimen (N=96) | Placebo (N=91)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Apallic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 21 (28) | 22 (25)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCT197 High Dose Regimen (N=92) | BCT197 Low Dose Regimen (N=96) | Placebo (N=91)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (2)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal vein occlusion (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Scleral hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 4 (6) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 3 (3)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 3 (4) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 4 (5) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 2 (4) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Blood potassium increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 3 (3) | 0 (0)
Gamma-glutamyltransferase abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Monocyte count increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Platelet count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein total decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (2) | 2 (3) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Apallic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1)
Hypotonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphoria (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 24 (33) | 32 (42) | 28 (41)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (5)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Paranasal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Tonsillar erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (5) | 2 (2) | 4 (4)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT02700919/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT02700919/SAP_001.pdf